CLINICAL TRIAL: NCT03213977
Title: A Multicenter,Randomized, Controlled (Comparative), Open, Prospective Study Evaluating an Efficacy of R-DA-EPOCH and R-CEOP90, With or Without Upfront Auto-HSCT，in Newly Diagnosed Young Patients With High-risk DLBCL
Brief Title: R-DA-EDOCH Versus R-CEOP90, With/Without Upfront Auto-HSCT in Young Patients With High-risk DLBCL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Jianda Hu, Prof., Fujian Medical University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: DLBCL-005
Record Dates: First submitted 2017-07-03; First posted 2017-07-11 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: DLBCL, R-DA-EPOCH, R-CEOP90, auto-HSCT
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Masking Description: Open Label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I:R-DA-EPOCH (Active Comparator): Protocol involves 6 cycles. Patients with complete remission or partial remission undergo auto-HSCT after 6 cycles.
  Interventions: Drug: R-DA-EPOCH
- Arm II:R-CEOP90 (Experimental): Protocol involves 6 cycles. Patients with complete remission or partial remission undergo auto-HSCT after 6 cycles.
  Interventions: Drug: R-CEOP90

INTERVENTIONS:
Drug: R-DA-EPOCH — R-DA-EPOCH-21 treatment for DLBCL patients between 16 to 60 years with high risk. Patients who meet the criteria for ASCT after reaching CR or PR will undergo ASCT, while those who do not meet the criteria or refuse to undergo ASCT, will continue with 2 cycles of immunochemotherapy.
  Arms: Arm I:R-DA-EPOCH
Drug: R-CEOP90 — R-CEOP90 treatment for DLBCL patients between 16 to 60 years with high risk. Patients who meet the criteria for ASCT after reaching CR or PR will undergo ASCT, while those who do not meet the criteria or refuse to undergo ASCT, will continue with 2 cycles of immunochemotherapy.
  Arms: Arm II:R-CEOP90

SUMMARY:
Patients initially are randomized into 2 arms:

Arm I: R-DA-EPOCH; Arm II: R-CEOP90;

Patients who achieved complete remission (CR) or partial remission (PR) after 6 cycles of R-DA-EPOCH (Arm I) or R-CEOP90 (Arm II), continue to have 2 more cycles for consolidation in each arm, or undergo stem cell harvest and auto-HSCT following standard institutional protocols.

DETAILED DESCRIPTION:
Patients initially are randomized into 2 arms:

Arm I: R-DA-EPOCH; Arm II: R-CEOP90;

Patients who achieved complete remission (CR) or partial remission (PR) after 6 cycles of R-DA-EPOCH (Arm I) or R-CEOP90 (Arm II), continue to have 2 more cycles for consolidation in each arm, or undergo stem cell harvest and auto-HSCT following standard institutional protocols.

The overall purpose of the study is to determine if R-CEOP90 followed by auto-HSCT has similar efficacy compared to that with R-DA-EPOCH.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-60 years
* Newly diagnosed DLBCL
* No previous treatment with chemotherapy and/or radiation therapy of DLBCL
* Presence of 2 or more signs of unfavorable prognosis: aaIPI≥2 or aaIPI=1 with Bulk (≥7.5cm)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy of ≥6 months
* Adequate hematological function
* Offer informed consent

Exclusion Criteria:

* Transformation of mature cell lymphomas in DLBCL
* Pretreated DLBCL
* HIV-associated DLBCL
* Concomitant other cancer
* Congestive heart failure, unstable angina, severe cardiac arrhythmias and conduction disturbances, myocardial infarction
* Renal insufficiency (serum creatinine greater than 0.2 mmol/L) (except cases with specific kidney infiltration, urinary tract compression by tumor conglomerate or presence of uric acid nephropathy due to massive cytolysis syndrome)
* Liver failure (except cases with liver tumor infiltration), acute hepatitis or active phase of chronic hepatitis B or C with serum bilirubin greater than 1.5 standards, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) greater than 3 standards, prothrombin index less than 70%
* Severe pneumonia (except cases with specific lungs infiltration), accompanied by respiratory failure (dyspnea > 30 in min., hypoxemia less than 70 mm Hg, when it is impossible to compensate situation in 2-3 days)
* Life-threatening bleeding (gastrointestinal, intracranial), with exception of bleeding due to tumor infiltration of organs (stomach, intestines, uterus, etc.) and disseminated intravascular coagulation due to underlying disease complications after their successful conservative treatment
* Severe mental disorders (delusions, severe depressive syndrome and other manifestations of productive symptoms) not related with specific infiltration of central nervous system
* Decompensated diabetes
* Pregnancy

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 475 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2024-07-13 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | Two-year survival
  Time to disease progression is calculated in months from day of enrollment in the study until disease progression, as appropriate

SECONDARY OUTCOMES:
complete response | 6 cycles
  (physical examination, standard blood tests, including assessment of LDH level, thoracic and abdominal computerized tomography (together with any other anatomic site, as clinically indicated), bone marrow biopsy in case of bone marrow involvement and 18F-fludeoxyglucose positron emission tomography (18FDG-PET) (not mandatory) in case of residual measurable disease at the end of the chemoimmunotherapy)
overall survival | Two-year survival
  Survival time is calculated in months from day of enrollment in the study until death, as appropriate
Incidence of Treatment-Emergent Adverse Events | During the treatment
  Adverse Events (AEs) occurring during the protocol-specified reporting period are documented.

CONTACTS AND LOCATIONS:
Overall Officials: Jianda Hu, Prof., Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China